CLINICAL TRIAL: NCT03561558
Title: Open, Randomized, Cross-over, Two Period, Two-sequence, One-center, Bioequivalence Study of Ibuprofen D, Oral Suspension, 200 mg / 5ml (Pharmtechnology, Belarus) and Nurofen® for Children, Oral Suspension 100 mg / 5 ml (Reckitt Benckiser Healthcare International Ltd, UK) in Healthy Volunteers Under Fasting Conditions
Brief Title: Bioequivalence Study of Ibuprofen D, Oral Suspension, 200 mg/5ml and Nurofen®, Oral Suspension 100 mg/5 ml in Healthy Volunteers Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmtechnology LLC (Industry)
Collaborators: ClinPharmInvest, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: FRM-03-IBU/21/11/17
Record Dates: First submitted 2018-06-07; First posted 2018-06-19 (Actual); Last update posted 2018-11-01 (Actual); Status verified 2018-06

CONDITIONS: Healthy
Keywords: Bioequivalence

STUDY DESIGN:
Masking Description: This study is an open label study; the subjects and the investigator will not be blinded towards the identity of the investigational products. However, analysts will be blinded towards identity of investigational products administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ibuprofen D, oral suspension (Experimental): Ibuprofen oral suspension, 200 mg/ 5 ml is the test product. In period 1 and period 2, 15 of 30 subjects will be given single oral dose (5 ml containing 200 mg of ibuprofen) of suspension.
  Interventions: Drug: Ibuprofen D
- Nurofen® for Children, oral suspension (Active Comparator): Nurofen® for Children oral suspension, 100 mg/ 5 ml is the reference product. In period 1 and period 2, 15 of 30 subjects will be given single oral dose (10 ml containing 200 mg of ibuprofen) of suspension.
  Interventions: Drug: Nurofen® for Children

INTERVENTIONS:
Drug: Ibuprofen D — Ibuprofen D, oral suspension, 200 mg / 5ml, manufactured by LLC Pharmtechnology, Belarus
  Arms: Ibuprofen D, oral suspension
Drug: Nurofen® for Children — Nurofen® for Children, Oral Suspension, 100 mg / 5 ml, marketed by Reckitt Benckiser Healthcare International Ltd, UK
  Arms: Nurofen® for Children, oral suspension

SUMMARY:
To demonstrate bioequivalence of single dose test formulation of Ibuprofen,oral suspension 200 mg/5 ml (containing ibuprofen 200 mg) of Pharmtechnology LLC, Republic of Belarus with reference Nurofen® for Children, oral suspension 100 mg / 5 ml (containing ibuprofen 100 mg) of "Reckitt Benckiser Healthcare International Ltd, .", UK in normal, healthy, adult, human subjects under fasting conditions.To monitor adverse events and ensure the safety

DETAILED DESCRIPTION:
Total 30 normal healthy adult subjects will be enrolled in the study. Subjects will be administered either the Test (5 ml of oral suspension containing 200 mg of ibuprofen) or the Reference Product (10ml of oral suspension containing 200 mg of ibuprofen) with 200 mL of water in each period as per the randomization schedule. Subjects will fast for at least 10 hours prior to administration of the study drugs and for four (4) hours after administration of the study drugs during each study period. Standardized meals will be provided in each study period. Water will not be accessible to the subjects 1 hour to administration of the study drugs and 2 hours after administration of the study drugs in each period. A total of 20 blood samples will be withdrawn for pharmacokinetic profiling during each study period. The plasma concentrations of R- and S-enantiomers of ibuprofen will be measured by a validated LC-MS/MS analytical method. ANOVA will be performed on log transformed pharmacokinetic parameters Cmax, AUC0-t and 90% confidence interval will be constructed for the ratio of geometric least square mean of the Test and Reference products, obtained from the log-transformed data. Bioequivalence will be concluded if the ratio estimate as well as its 90% confidence interval of S-enantiomers of ibuprofen, both falls within the acceptable range of 80.00% to 125.00% for Cmax, AUC0-t.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult human subjects, aged between 18 to 45 years.
2. Subjects with Body Mass Index (BMI) 18.5 to 30 kg/m2.
3. Female subjects with a negative pregnancy test.
4. Non-lactating females.
5. If subject is a female and is of child bearing potential, she should be practicing an acceptable non-hormonal method of birth control for the duration of the study(at least 14 days before the start of the study, throughout the study and 14 days after the completion of the study), such as a combination of male condom and diaphragm with spermicide.
6. If subject is a male and and has a female partner of child bearing potential, he should be practicing an acceptable method of birth control for the duration of the study(at least 14 days before the start of the study, throughout the study and 14 days after the completion of the study), such as a combination of male condom and spermicide (double barrier method).
7. Subjects having no clinically significant medical history and no clinically significant abnormalities in general physical examination, laboratory assessments, 12-lead ECG, chest X-Ray or vital signs.
8. Subjects are able to understand the requirements of the study, to sign a written informed consent, and also to accept all the restrictions imposed during the course of the study, and to agree to return for the required investigations.

Exclusion Criteria:

1. Subjects with a known history of allergic disorders.
2. Subjects with a known history of drug hypersensitivity to ibuprofen d or any excipients of the formulation.
3. Subjects with a known history of drug intolerance.
4. Subjects with history of psychiatric disorders.
5. Subjects with history of epilepsy, seizures, other neurological disorders.
6. Subjects on a low sodium diet for 2 weeks before the start study, or on any special diet (for example, vegetarian, vegan) or follow a special lifestyle (night shifts,extreme physical work).
7. Use of hormonal contraceptives either oral or implants within 6 months prior to first period dosing.
8. Female subjects of child bearing potential who have had an unprotected sexual intercourse with an unsterilized male sexual partner within 30 days before the start of the study
9. Use of any xanthine-containing food or beverages (tea, coffee, chocolates, soft drinks like cola, etc.) for at least 72 hours prior to the start of the study.
10. Use of citrus fruits (including grapefruit and grapefruit juice) and cranberries (including juices,etc.) for at least 14 days prior to the start of the study.
11. Subjects with a history of disorders of cardiovascular, bronchopulmonary, neuroendocrine system, and also the gastrointestinal tract, liver, kidney and blood.
12. Subjects with a history of other disorders that, at the discretion of the Principal Investigator, can affect absorption, distribution, metabolism or excretion of both drugs or increase the risk of adverse effects.
13. Subjects with a history of surgical interventions on the gastrointestinal tract except for appendectomy.
14. Subjects with a history acute infectious illnesses within 4 weeks prior to the start of the study.
15. Subjects with abnormalities in resting heart rate (>80 beats/min or <60 beats/min), blood pressure either hypotensive episode (systolic blood pressure <100 mmHg or diastolic blood pressure <70 mmHg) or hypertension (systolic blood pressure ≥ 130 mmHg or diastolic blood pressure ≥90 mmHg), in ECG
16. Use of known inhibitors or inducers of liver function, in particular isoenzyme CYP 3A4 (example of inducers: omeprazole, cimetidine, drugs, containing St. John's wort extract, barbiturates, carbamazepine, phenytoin, glucocorticoids; example of inhibitors: antiviral drugs, clarithromycin, ciprofloxacin, gestodene, etc.) within 2 months prior to the start of the study.
17. Use of any drugs with systemic absorption within14 days prior to the start of the study.
18. Use of OTC drugs, including herbs and nutritional supplements within 7 days prior to the Dosing Date. (including vitamins and natural food additives, phyto supplements,herbal preparations such as, cat's claw, angelica officinalis, oenothera, feverfew, garlic, ginger, ginkgo, red clover, horse chestnut, green tea, ginseng).
19. Depot injection or implants of any drugs within 3 months prior to the start of the study.
20. Donation of plasma or blood (450 ml or more) within 2 months prior to the start of the study.
21. Intake of more than 10 units alcohol per week (1 unit of alcohol is equivalent to ½ liter of beer, 200 ml dry wine or 50 ml of spirits) or history alcoholism, drug addiction, drug abuse.
22. Smoking more than 10 cigarettes per day.
23. Participation in other clinical trials of medicines within 3 months prior to the start of the study.
24. Positive test for syphilis, hepatitis B, hepatitis C or HIV.
25. Positive pregnancy test (for female subjects with child bearing potential).
26. Breast-feeding.
27. Positive test for alcohol.
28. Positive urinary screen test for drugs of abuse.
29. Subjects with a history of a rare hereditary intolerance to galactose and/or sucrose, a deficiency of lactase, glucose-galactose malabsorption syndrome.
30. Subjects with clinically significant abnormal laboratory values and results of imaging studies.
31. Subjects who refuse to comply with the study protocol and/or not credible therein and who are, at the discretion of the Principal Investigator, unable to understand and assess the information about the study, expected risks and possible discomfort in the process of signing written informed consent.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2018-06-24 (Actual); Study Completion 2018-06-25 (Actual)

PRIMARY OUTCOMES:
Primary pharmacokinetic parameter for S-enantiomer of ibuprofen | 8 days
  Peak Plasma Concentration (Cmax)
Primary pharmacokinetic parameter for S-enantiomer of ibuprofen | 8 days
  Area under the plasma concentration versus time curve from time 0 to the last measured concentration (AUC0-t)

SECONDARY OUTCOMES:
Safety and tolerability of the investigational products (testing and reference) | 22 days
  Number of adverse events, number of deaths, number of severe adverse events in subjects who have taken at least one dose of investigational products.
Secondary pharmacokinetic parameter for S-enantiomer of ibuprofen | 8 days
  Area under the plasma concentration versus time curve from time 0 to to infinite time(AUC0-∞)
Secondary pharmacokinetic parameter for S-enantiomer of ibuprofen | 8 days
  Time of maximum measured plasma concentration (Tmax)
Secondary pharmacokinetic parameter for S-enantiomer of ibuprofen | 8 days
  Elimination or terminal half-life (T1/2)
Secondary pharmacokinetic parameter for S-enantiomer of ibuprofen | 8 days
  Elimination rate constant (Kel)
Secondary pharmacokinetic parameter for S-enantiomer of ibuprofen | 8 days
  Residual area (AUCresid)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Khokhlov, Professor, Principal Investigator — ClinPharmInvest, LLC
Locations (1):
- State Autonomous Healthcare Facility of the Yaroslavl Region "Clinical Hospital No. 2", Yaroslavl, Yaroslavl Oblast, Russia

IPD SHARING:
Plan to Share IPD: Undecided
The Company may provide the individual participant data after privacy protection on case by case basis.